CLINICAL TRIAL: NCT00378469
Title: Study of the Effects of Muscular Activity on Iron Metabolism: A Pilot Study on Healthy Volunteers
Brief Title: Study of the Effects of Muscular Activity on Iron Metabolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rennes University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DGS 2006/0415; LOC/05-07; CIC0203/061
Record Dates: First submitted 2006-09-19; First posted 2006-09-20 (Estimated); Last update posted 2007-07-12 (Estimated); Status verified 2007-05

CONDITIONS: Iron Overload; Iron Deficiency
Keywords: Hepcidin; Hemojuvelin; Iron; Healthy volunteers
MeSH Terms: conditions — Iron Overload; Iron Deficiencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: 45 minute exercise on ergocycle

SUMMARY:
The aim of this study is to evaluate the effect of muscular exercise on iron metabolism in healthy volunteers. Fourteen healthy male subjects will have to pedal on an ergocycle for 45 minutes, and urine and blood samples will be collected regularly to measure hemojuvelin, hepcidin, iron and transferrin levels.

DETAILED DESCRIPTION:
Hemojuvelin has been described as interfering with hepcidin, a key regulator of iron homeostasis. Hemojuvelin is mainly produced by muscle, and the relationship between exercise and iron metabolism can be questioned about.

The aim of this study is to evaluate the effect of muscular exercise on iron metabolism in healthy volunteers. Fourteen healthy male subjects will be investigated at two periods according to a cross-over design after:

1. 45 minutes of exercise on the ergocycle; and
2. no physical exercise.

Urine and blood samples will be collected at both periods regularly to measure hemojuvelin, hepcidin, iron and transferrin levels.

ELIGIBILITY:
Inclusion Criteria:

* Male individuals aged between 18 and 40 years old
* Body mass index (BMI) between 18 and 25
* Normal at clinical examination
* Normal biological variables
* Written informed consent

Exclusion Criteria:

* Mutation C282Y of the HFE gene
* Iron metabolism abnormality
* Inflammatory syndrome
* Chronic pathology or ongoing treatment
* Tobacco smoking, alcohol consuming more than 30g/day
* History of transfusion or blood-giving within 3 months
* Positive serology for hepatitis B virus (HBV), hepatitis C virus (HCV) or HIV.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2006-09

PRIMARY OUTCOMES:
Pharmacokinetics of urinary hepcidin
Pharmacokinetics of blood hemojuvelin

SECONDARY OUTCOMES:
Pharmacokinetics of urine and blood iron, transferrin, interleukin-6 (IL-6) and ferritin

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Brissot, MD, Principal Investigator — Rennes University Hospital; Bruno Laviolle, MD, Study Chair — Rennes University Hospital
Locations (2):
- France (2):
  - Service des Maladies du Foie - Hôpital de Pontchaillou, Rennes
  - Unité de Biologie et Médecine du Sport - Hôpital de Pontchaillou, Rennes